CLINICAL TRIAL: NCT04103437
Title: Evaluation of Harmonicity in Running Gait by the Use of Innovative Techniques of Video Analysis: Effects on Metabolic Consumption and Running Injuries Risk
Brief Title: Evaluation of Harmonicity in Running Gait by the Use of Innovative Techniques of Video Analysis
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Microgate Srl (Unknown); Universita di Verona (Other)
Responsible Party: Sponsor
Other Study IDs: harmrun fdg
Record Dates: First submitted 2018-11-27; First posted 2019-09-25 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2018-10

CONDITIONS: Injuries
Keywords: running harmonicity; running related injuries
MeSH Terms: conditions — Wounds and Injuries | interventions — Metabolic Networks and Pathways; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- recreational runners: Recreational runners (minimum of 2 running session and 20km of total mileage per week), with seasonal best on half-marathon comprised between 1h20' and 2h00'. Age > 18 and < 60 years. Free from musculoskeletal injuries from at least three months.
  Interventions: Diagnostic Test: Maximal incremental running test; Diagnostic Test: Metabolic and movement analysis of running; Other: Questionnaires

INTERVENTIONS:
Diagnostic Test: Maximal incremental running test — Maximal incremental running test with measures of metabolic, spatio-temporal parameters and video recording with camera in the frontal plane.
  video recording of frontal view, metabolic and spatio-temporal measures of three (self-selected speed, + and - 20 percentage of self-selected speed) 6 minutes running test monthly (12 months) follow-up questionnaire
Diagnostic Test: Metabolic and movement analysis of running — Running analysis of three six minutes running test (self-selected speed, + and - 20% of the self-selected speed) by video recording with camera in the frontal plane, and acquisition of the metabolic and spatio-temporal parameters
Other: Questionnaires — Monthly follow-up questionnaire (12 months) about training habits and injuries

SUMMARY:
This study aims to demonstrate the use of a digital video analysis method to evaluate harmonicity of running gait, through an holistic approach.

Furthermore, it explores the association of running gait harmonicity with running velocity and level of training and with running injuries risk .

DETAILED DESCRIPTION:
Aetiology of running related injuries is reported to be multifactorial but still not fully understood. Factors that impede the understanding of the mechanisms and aetiology of injury are the traditional segmental approach to the analysis of running gait and the lack of prospective studies.

A more holistic approach to analysis of movement could permit a more in depth comprehension of the injured state, trough a changing of point of view. This holistic approach is based on the harmonic nature of running gait.

Despite the everyday use of the term "harmonicity" within sporting domains, methods to measure running gait harmonicity is a theme still vaguely explored.

Traditional methods evaluate the movement quality of the whole body based on the motion analysis of specific segments, that are supposed to sufficiently represent the entire body. The search for a method to analyse harmonicity of cyclic movements with a real holistic approach, is therefore still open.

With these aims, an innovative video analysis method has been proposed, based on the measure of the frequency variation of the pixel brightness in the digital video of a cyclic movement.

ELIGIBILITY:
Inclusion Criteria:

* at least one year of running practice
* minimum two day of running/week
* minimum 20 km running/week
* seasonal best on half marathon comprised between 1h20' and 2h00'
* experienced in treadmill running practice
* sport medical certificate

Exclusion Criteria:

* have suffered in the last three months of musculoskeletal disease
* regular practice of sport activities different from running
* acute or chronic osteoarticular diseases or, in general, other pathology limiting physical activities
* use of drugs altering physical activity performance (hypnotic, psychoactive, non-steroidal anti-inflammatory drugs e.g.).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: recreational runners
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2018-11-03 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Correlation between running related injuries (RRI) and running gait harmonicity | 1year
  Verify if RRI risk is correlated with measures of harmonicity derived from Graal software (registered during three six minutes running test at low, self-selected, high speed):
  • Number of pixel of the nine principal frequencies RRI are registered by follow-up questionnaires each month .

SECONDARY OUTCOMES:
Correlation between running gait harmonicity and spatio-temporal running parameters | 1 year
  The association of running gait harmonicity measures with contact time, flight time, stride length and cadence will be evaluated at each running velocity.
Correlation between running gait harmonicity and metabolic parameters | 1 year
  The association of running gait harmonicity measures with VO2max, ventilation, respiratory exchange ratio and hearth rate.
Correlation between running related injuries (RRI) and running gait harmonicity | 1 year
  Verify if RRI risk is correlated with measures of harmonicity derived from Graal software (registered during three six minutes running test at low, self-selected, high speed): Signal/noise ratio (ratio between values of the principal frequencies and noise)

CONTACTS AND LOCATIONS:
Overall Officials: Guido Pasquini, Bs, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi
Locations (1):
- IRCCS Don Carlo Gnocchi, Florence, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huijben B, van Schooten KS, van Dieen JH, Pijnappels M. The effect of walking speed on quality of gait in older adults. Gait Posture. 2018 Sep;65:112-116. doi: 10.1016/j.gaitpost.2018.07.004. Epub 2018 Jul 10. PMID 30558916
- [Result] Lindsay TR, Yaggie JA, McGregor SJ. Contributions of lower extremity kinematics to trunk accelerations during moderate treadmill running. J Neuroeng Rehabil. 2014 Dec 12;11:162. doi: 10.1186/1743-0003-11-162. PMID 25495782
- [Result] Buist I, Bredeweg SW, Lemmink KA, van Mechelen W, Diercks RL. Predictors of running-related injuries in novice runners enrolled in a systematic training program: a prospective cohort study. Am J Sports Med. 2010 Feb;38(2):273-80. doi: 10.1177/0363546509347985. Epub 2009 Dec 4. PMID 19966104
- [Result] Videbaek S, Bueno AM, Nielsen RO, Rasmussen S. Incidence of Running-Related Injuries Per 1000 h of running in Different Types of Runners: A Systematic Review and Meta-Analysis. Sports Med. 2015 Jul;45(7):1017-26. doi: 10.1007/s40279-015-0333-8. PMID 25951917
- [Result] van Gent RN, Siem D, van Middelkoop M, van Os AG, Bierma-Zeinstra SM, Koes BW. Incidence and determinants of lower extremity running injuries in long distance runners: a systematic review. Br J Sports Med. 2007 Aug;41(8):469-80; discussion 480. doi: 10.1136/bjsm.2006.033548. Epub 2007 May 1. PMID 17473005
- [Result] Hreljac A. Etiology, prevention, and early intervention of overuse injuries in runners: a biomechanical perspective. Phys Med Rehabil Clin N Am. 2005 Aug;16(3):651-67, vi. doi: 10.1016/j.pmr.2005.02.002. PMID 16005398
- [Result] Vannatta CN, Kernozek TW. Patellofemoral joint stress during running with alterations in foot strike pattern. Med Sci Sports Exerc. 2015 May;47(5):1001-8. doi: 10.1249/MSS.0000000000000503. PMID 25202853
- [Result] Teng HL, Powers CM. Sagittal plane trunk posture influences patellofemoral joint stress during running. J Orthop Sports Phys Ther. 2014 Oct;44(10):785-92. doi: 10.2519/jospt.2014.5249. Epub 2014 Aug 25. PMID 25155651
- [Result] Valenzuela KA, Lynn SK, Mikelson LR, Noffal GJ, Judelson DA. Effect of Acute Alterations in Foot Strike Patterns during Running on Sagittal Plane Lower Limb Kinematics and Kinetics. J Sports Sci Med. 2015 Mar 1;14(1):225-32. eCollection 2015 Mar. PMID 25729311
- [Result] Hamill J, Palmer C, Van Emmerik RE. Coordinative variability and overuse injury. Sports Med Arthrosc Rehabil Ther Technol. 2012 Nov 27;4(1):45. doi: 10.1186/1758-2555-4-45. PMID 23186012
- [Result] Kiely J, Collins DJ. Uniqueness of Human Running Coordination: The Integration of Modern and Ancient Evolutionary Innovations. Front Psychol. 2016 Apr 11;7:262. doi: 10.3389/fpsyg.2016.00262. eCollection 2016. PMID 27148098
- [Result] Bredeweg SW, Kluitenberg B, Bessem B, Buist I. Differences in kinetic variables between injured and noninjured novice runners: a prospective cohort study. J Sci Med Sport. 2013 May;16(3):205-10. doi: 10.1016/j.jsams.2012.08.002. Epub 2012 Aug 24. PMID 22921763
- [Result] Iosa M, Bini F, Marinozzi F, Fusco A, Morone G, Koch G, Martino Cinnera A, Bonni S, Paolucci S. Stability and Harmony of Gait in Patients with Subacute Stroke. J Med Biol Eng. 2016;36(5):635-643. doi: 10.1007/s40846-016-0178-0. Epub 2016 Oct 7. PMID 27853414
- [Result] Bellanca JL, Lowry KA, Vanswearingen JM, Brach JS, Redfern MS. Harmonic ratios: a quantification of step to step symmetry. J Biomech. 2013 Feb 22;46(4):828-31. doi: 10.1016/j.jbiomech.2012.12.008. Epub 2013 Jan 12. PMID 23317758
- [Result] Stefanyshyn DJ, Stergiou P, Lun VM, Meeuwisse WH, Worobets JT. Knee angular impulse as a predictor of patellofemoral pain in runners. Am J Sports Med. 2006 Nov;34(11):1844-51. doi: 10.1177/0363546506288753. Epub 2006 May 30. PMID 16735584